CLINICAL TRIAL: NCT06039787
Title: Effects of One Exercise Training Session on Brain Insulin Responsiveness
Brief Title: Exercise Training on Brain Insulin Responsiveness
Acronym: acEx
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 226/2023BO2
Record Dates: First submitted 2023-09-06; First posted 2023-09-15 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-09

CONDITIONS: Insulin Resistance; Obesity
Keywords: Exercise; functional magnetic resonance imaging; Intranasal insulin
MeSH Terms: conditions — Insulin Resistance; Obesity; Motor Activity

STUDY DESIGN:
Intervention Model Description: In a cross-over design, we will compare cerebral response from before to after intranasal insulin administration after a single bout of HIIT or MICT compared to a control condition without exercise.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- moderate intensity continuous training (Experimental)
  Interventions: Behavioral: single bout of moderate intensity continuous training (MICT)
- High-intensity interval training (Experimental)
  Interventions: Behavioral: single bout of High Intensity Interval Training (HIIT)
- Waiting condition (Placebo Comparator)
  Interventions: Behavioral: waiting control

INTERVENTIONS:
Behavioral: single bout of moderate intensity continuous training (MICT) — the MICT consists of 60 min continuous cycling
  Arms: moderate intensity continuous training
Behavioral: single bout of High Intensity Interval Training (HIIT) — HIIT consists of 10-min warm-up at the power output corresponding to 50% peak power output (PPO), 4 x 4-min intervals at a power output corresponding to 75% PPO with a 4-min active resting period at 30% PPO to recover
  Arms: High-intensity interval training
Behavioral: waiting control — sitting in a waiting room for 60 min
  Arms: Waiting condition

SUMMARY:
The overarching goal of the current study is to investigate the effect of one acute bout of exercise on the brain insulin responsiveness in a cross-over study design. To this end, investigators will compare the effect of two single endurance exercise sessions with different intensities, namely moderate intensity continuous training (MICT) and high-intensity-interval-training (HIIT), which will be performed in a randomized order. This will be compared to a waiting control condition.

DETAILED DESCRIPTION:
Investigate one acute bout of exercise on the brain insulin responsiveness using functional magnetic resonance imaging in combination with intranasal insulin in healthy participants of normal-weight and overweight/obesity. Two single endurance exercise sessions with different intensities will be evaluated, namely moderate intensity continuous training (MICT) and high-intensity interval training (HIIT). This will be compared to a waiting control condition. In a cross-over design, investigators will compare cerebral response from before to after intranasal insulin administration after a single bout of HIIT or MICT compared to a control condition without exercise. Cerebral response is defined as the cerebral blood flow and resting state functional connectivity in response to intranasal insulin. Secondary outcomes include changes in blood metabolites and proteins and changes in eating behavior.

ELIGIBILITY:
Inclusion Criteria:

* BMI between ≥ 19.5 to 39 kg/m2-
* Less than 150 min/week for moderate-intensity physical activity
* Less than 75 min/week for Vigorous- intensity exercise (WHO recommendations for regular physical activity of adults)
* Written consent to participate in the study
* Written consent to be informed about incidental findings

Exclusion Criteria

* Type 2 diabetes, cardiovascular diseases such as chronic heart failure, myocardial infarction, status post stroke
* Limitations to participate in ergometer-based exercise (balance and coordination disorders, orthopedic problems, …)
* Insufficient knowledge of the German language
* Persons who cannot legally give consent
* Pregnancy or lactation
* History of severe mental or somatic disorders including neurological diseases (incl. epileptic seizures and migraines)
* Taking psychotropic drugs
* Taking medications that influence glucose metabolism
* Regular use of analgesic drugs
* Taking anticoagulant agents
* Previous bariatric surgery
* Acute infection within the last 4 weeks
* Hemoglobin values less than 12g/dl for women, less than 14 g/dl for men
* Other diseases that in the opinion of the investigator may jeopardize the success of the study or indicate a risk to the volunteer
* Current participation in a lifestyle intervention study or a pharmaceutical study
* Metal implants which cannot be removed as pacemakers, artificial heart valve, electrical devices as insulin pumps, large tattoos, retainer over more than 4 teeth, contraceptive coil, implanted magnetic metal parts as screws or plates after a surgery
* Persons with claustrophobia
* Temperature-sensitive person
* Persons with tinnitus or increased sensitivity to loud sounds

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Cerebral response after intranasal insulin administration | 1 hour after exercise or waiting control
  The resting-state cerebral response from before to after intranasal insulin administration after a single bout of HIIT or MICT exercise compared to a control condition without exercise (i.e., waiting control)

SECONDARY OUTCOMES:
Task based brain activation after high-intensity-interval-training (HITT) or moderate intensity continuous training (MICT) compared to control condition | 1 hour after exercise or waiting control
  Food cue reactivity after a single bout of HIIT or MICT exercise compared to a control condition without exercise (i.e., waiting control)
Subjective feeling of hunger and food craving | baseline, 1 hour after breakfast, 1 hour, 2 hour, 3 hours after exercise or waiting control
  Questionnaire assessment before and after exercise or waiting control.
Changes in Blood-brain barrier integrity | 1 hour after exercise or waiting control
  Robust multiple echo-time arterial spin labelling based Blood Brain Barrier integrity measurements from before to after intranasal insulin administration after a single bout of HIIT or MICT exercise compared to a control condition without exercise (i.e., waiting control)
Performance during cognitive tasks | 1 hour after exercise or waiting control
  Cambridge Cognition Tests Battery to assess memory and inhibitory control using the paired associates learning task, the pattern recognition memory task and the stop-signal reaction task.
Changes in exerkines from plasma samples | baseline, 1 hour after breakfast, 1 hour, 2 hour, 3 hours after exercise or waiting control
  Blood sampling at 5 time points before and after a single bout of HIIT or MICT exercise compared to a control condition without exercise (i.e., waiting control)
Change in incretins from plasma samples | baseline, 1 hour after breakfast, 1 hour, 2 hour, 3 hours after exercise or waiting control
  Blood sampling at 5 time points before and after a single bout of HIIT or MICT exercise compared to a control condition without exercise (i.e., waiting control)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas L. Birkenfeld, MD, Study Director — Institute for Diabetes research and Metabolic Diseases at the University of Tubingen
Locations (1):
- University Clinic Tübingen, Department of Internal Medicine IV, Tübingen, Germany